CLINICAL TRIAL: NCT05879419
Title: Efficacy, Immunogenicity and Safety of Recombinant Vaccine Against Herpes Zoster (RZV or SHINGRIX®) in Patients With Autoimmune Rheumatic Diseases
Brief Title: Recombinant Herpes Zoster Vaccine in Patients With Autoimmune Rheumatic Diseases
Acronym: RZVRheum
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 67374823.0.0000.0068
Record Dates: First submitted 2023-05-02; First posted 2023-05-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis; Spondylitis, Ankylosing; Spondyloarthritis; Systemic Lupus Erythematosus; Sjogren's Syndrome; Systemic Sclerosis; Idiopathic Inflammatory Myopathies; Vasculitis, Systemic; Juvenile Idiopathic Arthritis; Dermatomyositis, Juvenile; Behçet Disease
Keywords: Recombinant herpes zoster vaccine; Herpes zoster; Autoimmune rheumatic diseases; Disease activity; Safety; Immunogenicity; Disease-modifying anti-rheumatic drugs; Biological disease-modifying anti-rheumatic drugs; Glucocorticoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Spondylarthritis; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Systemic; Myositis; Systemic Vasculitis; Arthritis, Juvenile; Dermatomyositis; Behcet Syndrome; Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Subproject A: Randomized prospective study of adult patients with ARDs who will receive two intramuscular doses of RZV 6 weeks apart or placebo.
  Subproject B: Specific studies will evaluate the effect of drug withdrawal (MTX and MMF) after vaccination in increasing the immune response in patients with ARDs with controlled baseline disease. Randomization of patients with ARDs with well-controlled disease selected for the MTX discontinuation protocol will divide them into two groups: MTX-suspension, in which MTX will be suspended for 2 weeks after each vaccine dose, and another group that will maintain stable therapy (MTX-maintenance), with assessments of immunogenicity and disease activity. The same applies to patients undergoing the MMF discontinuation protocol (but the MMF suspension time will be one week after each vaccine dose).
Who Masked: Participant, Investigator
Masking Description: Subproject A: Randomized prospective study of adult patients with ARDs who will receive two intramuscular doses of RZV 6 weeks apart or placebo.
  Subproject B: Specific studies will to evaluate the effect of drug withdrawal (MTX and MMF) after vaccination in increasing the immune response in patients with ARDs with controlled baseline disease. Randomization of patients with ARDs with well-controlled disease selected for the MTX discontinuation protocol will divide them into two groups: MTX-suspension, in which MTX will be suspended for 2 weeks after each vaccine dose, and another group that will maintain stable therapy (MTX-maintenance).
  The same applies to patients undergoing the MMF discontinuation protocol (but the MMF suspension time will be one week after each vaccine dose).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Subproject A: Patients with ARDs who received the vaccine at study entry (P1) (Active Comparator): Patients with ARDs who received the vaccine at study entry (P1) (n = 590). ARD patients will be randomly assigned in a 1:1 ratio, with the use of an automated Web and telephone system, to one of two subgroups: P1, patients allocated to receive vaccine right after randomization (at D0 and D42), and P2, patients allocated to receive placebo at D0 and D42. Subsequently, blindness will be broken at D84 and P2 patients will receive vaccine doses at the D84 and D126.
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV)
- Subproject A: Patients with ARDs who received the placebo at study entry (P2) (Placebo Comparator): Subproject A: Patients with ARDs who received the placebo at study entry (P2) (n = 590).
  ARD patients will be randomly assigned in a 1:1 ratio, with the use of an automated Web and telephone system, to one of two subgroups: P1, patients allocated to receive vaccine right after randomization (at D0 and D42), and P2, patients allocated to receive placebo at D0 and D42. Subsequently, blindness will be broken at D84 and P2 patients will receive vaccine doses at the D84 and D126.
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV); Other: Placebo
- Subproject A: Control group of non-immunosuppressed individuals (CG) (Active Comparator): Subproject A: Control group of non-immunosuppressed individuals (CG) (n = 393). The control group of non-immunosuppressed individuals (CG) (≥50 years old) will be invited to receive the vaccine at study entry (3 patients:1 control).
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV)
- Subproject B: MTX-withhold (Active Comparator): Subproject B: MTX-withhold (n = 101). Patients using MTX at a stable dose for at least 12 weeks, prednisone maximum dose of 5 mg/day, in association or not with other drugs except rituximab, to be randomized into two arms: one that will withhold MTX for 2 weeks after each vaccine dose (MTX-withhold) and other that will maintain stable therapy (MTX-maintain).
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV); Other: MTX Discontinuation
- Subproject B: MTX-maintain (Active Comparator): Subproject B: MTX-maintain (n = 101). Patients using MTX at a stable dose for at least 12 weeks, prednisone maximum dose of 5 mg/day, in association or not with other drugs except rituximab, to be randomized into two arms: one that will withhold MTX for 2 weeks after each vaccine dose (MTX-withhold) and other that will maintain stable therapy (MTX-maintain).
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV); Other: MTX maintain
- Subproject B: MMF-withhold (Active Comparator): Subproject B: MMF-withhold (n = 115). Patients with ARDs using MMF at a stable dose for at least 12 weeks, prednisone maximum dose of 7.5 mg/day, not associated with other immunosuppressive therapy, will be consecutively evaluated at outpatient clinics regarding disease activity. Those considered to be at stable disease (at remission or low disease activity according to specific standardized disease activity indexes) will be randomized (1:1) into two arms: one that will withhold MMF for one week after each vaccine dose (MMF-withhold) and other that will maintain stable therapy (MMF-maintain).
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV); Other: MMF Discontinuation
- Subproject B: MMF-maintain (Active Comparator): Subproject B: MMF-maintain (n = 115). Patients with ARDs using MMF at a stable dose for at least 12 weeks, prednisone maximum dose of 7.5 mg/day, not associated with other immunosuppressive therapy, will be consecutively evaluated at outpatient clinics regarding disease activity. Those considered to be at stable disease (at remission or low disease activity according to specific standardized disease activity indexes) will be randomized (1:1) into two arms: one that will withhold MMF for one week after each vaccine dose (MMF-withhold) and other that will maintain stable therapy (MMF-maintain).
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (RZV); Other: MMF maintain

INTERVENTIONS:
Biological: Recombinant Herpes Zoster Vaccine (RZV) — RZV comprise 50 μg of recombinant VZV glycoprotein E and the liposome-based AS01B adjuvant system (which contains 50 μg of 3-O-desacyl-4'-monophosphoryl lipid A [MPL] and 50 μg of Quillaja saponaria Molina, fraction 21 (QS21, licensed by GSK from Antigenics, a subsidiary of Agenus)). Vaccine will be administered (0.5 ml) into the deltoid muscle at inclusion and 6 weeks (two doses).
  Other Names: Shingrix®
Other: MTX Discontinuation — Evaluation of discontinuation of the use of methotrexate (MTX) for 2 weeks after each vaccine dose in ARD patients: patients using MTX at a stable dose for at least 12 weeks, prednisone maximum dose of 5 mg/day, in association or not with other drugs except rituximab will be consecutively evaluated at outpatient clinics regarding disease activity. Those considered to be at stable disease (at remission or low disease activity according to specific standardized disease activity indexes) will be randomized (1:1) into two arms: one that will withhold MTX for 2 weeks after each vaccine dose (MTX-withhold) and other that will maintain stable therapy (MTX-maintain).
  Arms: Subproject B: MTX-withhold
Other: MMF Discontinuation — Evaluation of discontinuation of the use of mycophenolate mofetil (MMF) for one week after each vaccine dose in ARD patients: patients using MMF at a stable dose for at least 12 weeks, prednisone maximum dose of 7.5 mg/day, not associated with other immunosuppressive therapy, will be consecutively evaluated at outpatient clinics regarding disease activity. Those considered to be at stable disease (at remission or low disease activity according to specific standardized disease activity indexes) will be randomized (1:1) into two arms: one that will withhold MMF for 2 weeks after each vaccine dose (MMF-withhold) and other that will maintain stable therapy (MMF-maintain).
  Arms: Subproject B: MMF-withhold
Other: Placebo — Patients with ARDs who received the placebo at study entry (P2). ARD patients will be randomly assigned in a 1:1 ratio, with the use of an automated Web and telephone system, to one of two subgroups: P1, patients allocated to receive vaccine right after randomization (at D0 and D42), and P2, patients allocated to receive placebo at D0 and D42. Subsequently, blindness will be broken at D84 and P2 patients will receive vaccine doses at the D84 and D126.
  Arms: Subproject A: Patients with ARDs who received the placebo at study entry (P2)
Other: MTX maintain — MTX dose will be held stable after the two vaccine doses for comparison of vaccine immunogenicity and disease activity with the MTX-withhold group.
  Arms: Subproject B: MTX-maintain
Other: MMF maintain — MMF dose will be held stable after the two vaccine doses for comparison of vaccine immunogenicity and disease activity with the MMF-withhold group.
  Arms: Subproject B: MMF-maintain

SUMMARY:
Introduction: Patients with autoimmune rheumatic diseases (ARDs), rheumatoid arthritis (RA), juvenile idiopathic arthritis (JIA), psoriatic arthritis (PAs), ankylosing spondylitis (AS), systemic lupus erythematosus (SLE), primary Sjögren's syndrome (pSS) , systemic sclerosis (SSc), idiopathic inflammatory myopathies (IIM) and primary vasculitides, have a high risk of herpes zoster (HZ) infection. This increased susceptibility is caused by a deficient cell-mediated immune response due to the underlying disease and glucocorticoid and immunosuppressive treatments that impair the T-cell response, including conventional and unconventional synthetic disease-modifying anti-rheumatic drugs (DMARDs) and biological agents. In this context, the recent availability of a recombinant vaccine against HZ (RZV or Shingrix®), composed of recombinant VZV glycoprotein E (gE) and the AS01B adjuvant system (HZ/su), is a major progress regarding safety for immunosuppressed patients. Its effectiveness, however, has been clearly demonstrated for non-immunosuppressed patients and in selected populations of immunocompromised individuals. There are no prospective controlled studies evaluating the immunogenicity of RZV and its impact on the activity of the underlying disease, as well as its safety in patients with ARDs at high-risk for HZ.

Hypothesis: RZV has a good safety profile, including with respect to underlying rheumatic disease activity, in patients with ARDs at high risk of HZ.

Objectives: Primary: To assess the short-term safety profile in relation to underlying disease activity in patients with ARDs at high risk of HZ immunized with RZV compared to unvaccinated patients. Secondary: To evaluate the general safety of the vaccine in patients with ARDs at high risk of HZ immunized with RZV and non-immunosuppressed control subjects (CG); the humoral and cellular immunogenicity of RZV in patients with ARDs at high risk of HZ compared to CG; the influence of disease treatment on vaccine response; the 12-month persistence of humoral immunogenicity and incident cases of HZ. Specific studies will also be carried out to evaluate the effect of drug withdrawal (methotrexate-MTX and mycophenolate mofetil-MMF) after vaccination in increasing the immune response in patients with ARDs with controlled underlying disease.

On November 19, 2025, the institutional Ethics Committee approved an amendment to extend the project's timeframe to evaluate the following hypothesis:

- Immunosuppression may hamper 5-year long-term sustainability of humoral and cellular immune responses to RZV in ARD patients.

No new patients will be recruited, nor will any new intervations be performed. ARD patients previously included in the study and non-immunosuppressed control subjects who received both vaccine doses and collected samples for immunogenicity 6 weeks and one year after the second dose will be part of the proposed extension. A total of 1,025 ARD patients enrolled and 365 healthy controls will be included in the long-term follow-up phase. Considering a conservative 10% dropout, the final patient sample will be approximately 1,000.

Ethical statement: The extension protocol was approved by the institutional Ethics Committee (report 7.988.896), and written consent will be obtained from all participants prior to inclusion. Humoral immunogenicity will be evaluated by analyzing the serum concentrations of anti-gE antibodies (ELISA) of blood samples collected from participants at 5-year after complete VZR vaccination, as previously described (Cunningham et al., 2018). Cellular immunogenicity will be evaluated in a convenience sample (20% of the total research participants) of patients with ARDs and healthy controls at 5-year after complete VZR vaccination. Vaccine efficacy will be evaluated by incident cases of HZ in the period of 5 years after RZV vaccination. Participants will be followed for 5 years after the second RZV dose through monthly contacts and routine clinical visits every 3-6 months.

DETAILED DESCRIPTION:
Methods:

Subproject A: This is a phase 4 randomized prospective study of adult patients with ARDs who will receive two intramuscular doses of RZV 6 weeks apart. A control group of non-immunosuppressed individuals (CG) aged ≥ 50 years will also be included, in the proportion of 3 patients:1 control. Patients with ARDs will be randomly allocated into two groups: P1 and P2. CG and P1 will receive the vaccine soon after randomization, on D0 and D42. P2 will be vaccinated 12 weeks after randomization, on D84 and D126. All groups will collect blood samples immediately before vaccination, at baseline, and then receive the 1st dose of vaccine on the same day (D0 for CG and P1, and D84 for P2). The second dose will be applied 6 weeks after the first dose (D42 for P1 and CG, and D126 for P2). Blood samples for disease activity and immunogenicity will be collected 6 weeks after the 2nd dose (D84 for CG and P1 and D168 for P2). The influence of vaccination on disease activity will be evaluated in the first three months of follow-up through disease-specific activity indices. Safety analysis regarding adverse effects (AEs) of the vaccine will be performed using standardized questionnaires on D42 and D84 for CG and P1 and on D126 and D168 for P2. Severe AEs and incident cases of HZ will be evaluated throughout the study period. The persistence of immunogenicity will be evaluated one year after the 2nd dose (D407 for CG and P1, and D491 for P2).

Subproject B: Specific studies will also be carried out to evaluate the effect of drug withdrawal (MTX and MMF) after vaccination in increasing the immune response in patients with ARDs with controlled baseline disease. Randomization of patients with ARDs with well-controlled disease selected for the MTX discontinuation protocol will divide them into two groups: MTX-suspension, in which MTX will be suspended for 2 weeks after each vaccine dose, and another group that will maintain stable therapy (MTX-maintenance), with assessments of immunogenicity and disease activity. The same applies to patients undergoing the MMF discontinuation protocol (but the MMF suspension time will be one week after each vaccine dose). Based on a recently published study (Petri et al., 2023), discontinuation time of the MMF after each vaccine dose was reduced from two weeks to one week. In fact, these authors observed in a cohort of 334 patients with systemic lupus erythematosus that discontinuing MMF for one week after vaccination against COVID-19 (mRNA vaccine) improved vaccine efficacy without leading to exacerbations of the underlying disease (Petri et al., 2023). Thus, we considered it appropriate to reduce the MMF discontinuation time to one week after each dose of the recombinant vaccine for herpes zoster in our population of patients with autoimmune rheumatic diseases.

Total population: The total population will consist of 2005 participants comprising 1180 patients with ARDs (590 in P1 and 590 in P2), 393 healthy controls. 202 patients on the MTX maintenance/discontinuation RA protocol for two weeks after each vaccine dose, and 230 patients with ARDs on the MMF maintenance/discontinuation protocol for one week after each vaccine dose.

Immunogenicity analysis: Humoral immunogenicity will be evaluated through serum concentrations of anti-gE antibodies [enzyme-linked immunosorbent assay (ELISA)] of blood samples collected from participants pre-vaccination, 2 months and one year after the second dose of RZV. The frequencies of gE-specific CD4[2+] T cells will be measured after in vitro stimulation with a pool of peptides covering the gE ectodomain, by intracellular cytokine staining and detection by flow cytometry, in a convenience sample (20% of the total number of participants) from patients with ARDs and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be adults (≥18 years-old).
* ARD patients will be selected from patients regularly followed up at the Outpatient Rheumatology Clinics of the Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de São Paulo, São Paulo, SP, Brazil, according to the specific classification criteria: RA (Aletaha et al., 2010), SLE (Petri et al., 2012), pSS (Vitali et al., 2002), SSc (van den Hoogen et al., 2013), IIM (Lundberg et al., 2017), axial spondyloarthritis (axSpA) (Rudwaleit et al., 2009), PsA (Tillett et al., 2012) and granulomatosis with polyangiitis (Leavitt et al., 1990).
* Patients must be under current use of cyclophosphamide, mycophenolate mofetil, azathioprine, cyclosporin, tacrolimus, leflunomide, glucocorticoids, methotrexate, biologic therapy or JAKi with or without csDMARDs for at least one month prior to study inclusion.

Exclusion Criteria:

* history of any reaction or hypersensitivity to any component of the vaccine;
* previous HZ vaccination;
* any occurrence of Guillain-Barré syndrome;
* hospitalization, acute infectious disease or fever at the time of vaccination;
* pregnancy or lactation at the time of vaccination;
* history of HZ within the 12 months preceding the first dose of study vaccine;
* people living with HIV/AIDS (PLWHA).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2005 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Subproject A: Disease safety (flare) in ARD patients immunized with RZV in comparison to non-vaccinated ARD patients (placebo group) | Six months
  Flare will be defined as a new flare or worsening of previous disease activity according to established scores for each ARD or the change of therapy. Disease activity will be evaluated in ARD patients according to specific standardized disease activity indexes: RA (DAS28 - Disease Activity Score 28, RA-CDAI - Rheumatoid Arthritis Clinical Disease Activity Index), SLE (SLEDAI2K - Systemic Lupus Erythematosus Disease Activity Index 2000), pSS (ESSDAI- EULAR Sjögren's Syndrome Disease Activity Index), IIM (MMT - Manual Muscle Test), AxS (ASDAS - Ankylosing Spondylitis Disease Activity Score), and vasculitis (Birmingham Vasculitis Activity Score).
Subproject B: Effect of MTX discontinuation on immunogenicity in comparison to MTX maintenance | One year
  Humoral immunogenicity will be assessed through serum anti-gE antibody concentrations analysis (ELISA) of blood samples collected from participants at pre-vaccination, 6 weeks, and one-year after the second dose of RZV.
  The frequencies of gE-specific CD4[2+] T cells (CD4+ T-cells expressing at least 2 activation markers of the 4 markers assessed: interferon-γ, interleukin 2, tumor necrosis factor-α, and CD40 ligand) will be measured after in vitro stimulation with a pool of peptides covering the gE ectodomain, by intracellular cytokine staining and detection by flow cytometry, in a convenience sample (20% of total research participants).
Subproject B: Effect of MMF discontinuation on immunogenicity in comparison to MMF maintenance | One year
  Humoral immunogenicity will be assessed through serum anti-gE antibody concentrations analysis (ELISA) of blood samples collected from participants at pre-vaccination, 6 weeks, and one-year after the second dose of RZV.
  The frequencies of gE-specific CD4[2+] T cells (CD4+ T-cells expressing at least 2 activation markers of the 4 markers assessed: interferon-γ, interleukin 2, tumor necrosis factor-α, and CD40 ligand) will be measured after in vitro stimulation with a pool of peptides covering the gE ectodomain, by intracellular cytokine staining and detection by flow cytometry, in a convenience sample (20% of total research participants).

SECONDARY OUTCOMES:
Subproject A: Incidence of vaccine adverse events [safety and tolerability] in ARD patients immunized with RZV in comparison to non-vaccinated ARD patients (placebo group) and non-immunosupressed controls (control group) | Eighteen months
  A standardized diary card of AEs for recording of solicited local and systemic manifestations will be systematically provided to all patients and healthy controls collected for 7 days post each vaccination. Unsolicited AEs will be recorded within 6 weeks post each vaccination. Serious AEs (SAEs) and adverse events of special interest (AESIs) [potential immune mediated disorder (pIMDs)] will be evaluated throughout the entire study duration.
Subproject A: Humoral immunogenicity of the RZV in ARD patients in comparison to non-immunosupressed control group | One year
  Humoral immunogenicity will be assessed through serum anti-gE antibody concentrations analysis (ELISA) of blood samples collected from participants at pre-vaccination, 6 weeks, and one-year after the second dose of RZV.
  The frequencies of gE-specific CD4[2+] T cells (CD4+ T-cells expressing at least 2 activation markers of the 4 markers assessed: interferon-γ, interleukin 2, tumor necrosis factor-α, and CD40 ligand) will be measured after in vitro stimulation with a pool of peptides covering the gE ectodomain, by intracellular cytokine staining and detection by flow cytometry, in a convenience sample (20% of total research participants).

OTHER OUTCOMES:
Subproject A: Incident cases of HZ after RZV vaccination in ARD patients and in the non-immunosupressed control group | Eighteen months
  A suspected case of HZ will be defined as (1) a new unilateral, dermatomal, rash with pain (broadly defined to include allodynia, pruritus, or other abnormal sensations) without any alternative diagnosis or (2A) or a vesicular rash suggestive of varicella zoster virus infection regardless of the distribution, and no alternative diagnosis; without any alternative diagnosis. For each suspected case, the rash will be photographed and samples will be collected from three lesions to confirm the diagnosis of HZ by real-time polymerase-chain reaction (PCR) assay. If the PCR results were indeterminate or if samples were not available, the final diagnosis will be determined by unanimous agreement among the five members of an ascertainment committee, which includes a dermatologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abhishek A, Boyton RJ, Peckham N, McKnight A, Coates LC, Bluett J, Barber V, Cureton L, Francis A, Appelbe D, Eldridge L, Julier P, Valdes AM, Brooks T, Rombach I, Altmann DM, Nguyen-Van-Tam JS, Williams HC, Cook JA; VROOM study investigators. Effect of a 2-week interruption in methotrexate treatment versus continued treatment on COVID-19 booster vaccine immunity in adults with inflammatory conditions (VROOM study): a randomised, open label, superiority trial. Lancet Respir Med. 2022 Sep;10(9):840-850. doi: 10.1016/S2213-2600(22)00186-2. Epub 2022 Jun 27. PMID 35772416
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Anderson JK, Zimmerman L, Caplan L, Michaud K. Measures of rheumatoid arthritis disease activity: Patient (PtGA) and Provider (PrGA) Global Assessment of Disease Activity, Disease Activity Score (DAS) and Disease Activity Score with 28-Joint Counts (DAS28), Simplified Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI), Patient Activity Score (PAS) and Patient Activity Score-II (PASII), Routine Assessment of Patient Index Data (RAPID), Rheumatoid Arthritis Disease Activity Index (RADAI) and Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5), Chronic Arthritis Systemic Index (CASI), Patient-Based Disease Activity Score With ESR (PDAS1) and Patient-Based Disease Activity Score without ESR (PDAS2), and Mean Overall Index for Rheumatoid Arthritis (MOI-RA). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S14-36. doi: 10.1002/acr.20621. No abstract available. PMID 22588741
- [Background] Bastidas A, de la Serna J, El Idrissi M, Oostvogels L, Quittet P, Lopez-Jimenez J, Vural F, Pohlreich D, Zuckerman T, Issa NC, Gaidano G, Lee JJ, Abhyankar S, Solano C, Perez de Oteyza J, Satlin MJ, Schwartz S, Campins M, Rocci A, Vallejo Llamas C, Lee DG, Tan SM, Johnston AM, Grigg A, Boeckh MJ, Campora L, Lopez-Fauqued M, Heineman TC, Stadtmauer EA, Sullivan KM; ZOE-HSCT Study Group Collaborators. Effect of Recombinant Zoster Vaccine on Incidence of Herpes Zoster After Autologous Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2019 Jul 9;322(2):123-133. doi: 10.1001/jama.2019.9053. PMID 31287523
- [Background] Berkowitz EM, Moyle G, Stellbrink HJ, Schurmann D, Kegg S, Stoll M, El Idrissi M, Oostvogels L, Heineman TC; Zoster-015 HZ/su Study Group. Safety and immunogenicity of an adjuvanted herpes zoster subunit candidate vaccine in HIV-infected adults: a phase 1/2a randomized, placebo-controlled study. J Infect Dis. 2015 Apr 15;211(8):1279-87. doi: 10.1093/infdis/jiu606. Epub 2014 Nov 3. PMID 25371534
- [Background] Braun-Moscovici Y, Kaplan M, Braun M, Markovits D, Giryes S, Toledano K, Tavor Y, Dolnikov K, Balbir-Gurman A. Disease activity and humoral response in patients with inflammatory rheumatic diseases after two doses of the Pfizer mRNA vaccine against SARS-CoV-2. Ann Rheum Dis. 2021 Oct;80(10):1317-1321. doi: 10.1136/annrheumdis-2021-220503. Epub 2021 Jun 18. PMID 34144967
- [Background] Cunningham AL, Heineman TC, Lal H, Godeaux O, Chlibek R, Hwang SJ, McElhaney JE, Vesikari T, Andrews C, Choi WS, Esen M, Ikematsu H, Choma MK, Pauksens K, Ravault S, Salaun B, Schwarz TF, Smetana J, Abeele CV, Van den Steen P, Vastiau I, Weckx LY, Levin MJ; ZOE-50/70 Study Group. Immune Responses to a Recombinant Glycoprotein E Herpes Zoster Vaccine in Adults Aged 50 Years or Older. J Infect Dis. 2018 May 5;217(11):1750-1760. doi: 10.1093/infdis/jiy095. PMID 29529222
- [Background] Dagnew AF, Ilhan O, Lee WS, Woszczyk D, Kwak JY, Bowcock S, Sohn SK, Rodriguez Macias G, Chiou TJ, Quiel D, Aoun M, Navarro Matilla MB, de la Serna J, Milliken S, Murphy J, McNeil SA, Salaun B, Di Paolo E, Campora L, Lopez-Fauqued M, El Idrissi M, Schuind A, Heineman TC, Van den Steen P, Oostvogels L; Zoster-039 study group. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine in adults with haematological malignancies: a phase 3, randomised, clinical trial and post-hoc efficacy analysis. Lancet Infect Dis. 2019 Sep;19(9):988-1000. doi: 10.1016/S1473-3099(19)30163-X. Epub 2019 Aug 6. PMID 31399377
- [Background] Furer V, Eviatar T, Zisman D, Peleg H, Paran D, Levartovsky D, Zisapel M, Elalouf O, Kaufman I, Meidan R, Broyde A, Polachek A, Wollman J, Litinsky I, Meridor K, Nochomovitz H, Silberman A, Rosenberg D, Feld J, Haddad A, Gazzit T, Elias M, Higazi N, Kharouf F, Shefer G, Sharon O, Pel S, Nevo S, Elkayam O. Immunogenicity and safety of the BNT162b2 mRNA COVID-19 vaccine in adult patients with autoimmune inflammatory rheumatic diseases and in the general population: a multicentre study. Ann Rheum Dis. 2021 Oct;80(10):1330-1338. doi: 10.1136/annrheumdis-2021-220647. Epub 2021 Jun 14. PMID 34127481
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Lal H, Cunningham AL, Godeaux O, Chlibek R, Diez-Domingo J, Hwang SJ, Levin MJ, McElhaney JE, Poder A, Puig-Barbera J, Vesikari T, Watanabe D, Weckx L, Zahaf T, Heineman TC; ZOE-50 Study Group. Efficacy of an adjuvanted herpes zoster subunit vaccine in older adults. N Engl J Med. 2015 May 28;372(22):2087-96. doi: 10.1056/NEJMoa1501184. Epub 2015 Apr 28. PMID 25916341
- [Background] Leavitt RY, Fauci AS, Bloch DA, Michel BA, Hunder GG, Arend WP, Calabrese LH, Fries JF, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Wegener's granulomatosis. Arthritis Rheum. 1990 Aug;33(8):1101-7. doi: 10.1002/art.1780330807. PMID 2202308
- [Background] Lukas C, Landewe R, Sieper J, Dougados M, Davis J, Braun J, van der Linden S, van der Heijde D; Assessment of SpondyloArthritis international Society. Development of an ASAS-endorsed disease activity score (ASDAS) in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Jan;68(1):18-24. doi: 10.1136/ard.2008.094870. Epub 2008 Jul 14. PMID 18625618
- [Background] Lundberg IE, Tjarnlund A, Bottai M, Werth VP, Pilkington C, Visser M, Alfredsson L, Amato AA, Barohn RJ, Liang MH, Singh JA, Aggarwal R, Arnardottir S, Chinoy H, Cooper RG, Danko K, Dimachkie MM, Feldman BM, Torre IG, Gordon P, Hayashi T, Katz JD, Kohsaka H, Lachenbruch PA, Lang BA, Li Y, Oddis CV, Olesinska M, Reed AM, Rutkowska-Sak L, Sanner H, Selva-O'Callaghan A, Song YW, Vencovsky J, Ytterberg SR, Miller FW, Rider LG; International Myositis Classification Criteria Project consortium, The Euromyositis register and The Juvenile Dermatomyositis Cohort Biomarker Study and Repository (JDRG) (UK and Ireland). 2017 European League Against Rheumatism/American College of Rheumatology classification criteria for adult and juvenile idiopathic inflammatory myopathies and their major subgroups. Ann Rheum Dis. 2017 Dec;76(12):1955-1964. doi: 10.1136/annrheumdis-2017-211468. Epub 2017 Oct 27. PMID 29079590
- [Background] Medeiros-Ribeiro AC, Aikawa NE, Saad CGS, Yuki EFN, Pedrosa T, Fusco SRG, Rojo PT, Pereira RMR, Shinjo SK, Andrade DCO, Sampaio-Barros PD, Ribeiro CT, Deveza GBH, Martins VAO, Silva CA, Lopes MH, Duarte AJS, Antonangelo L, Sabino EC, Kallas EG, Pasoto SG, Bonfa E. Immunogenicity and safety of the CoronaVac inactivated vaccine in patients with autoimmune rheumatic diseases: a phase 4 trial. Nat Med. 2021 Oct;27(10):1744-1751. doi: 10.1038/s41591-021-01469-5. Epub 2021 Jul 30. PMID 34331051
- [Background] Mukhtyar C, Lee R, Brown D, Carruthers D, Dasgupta B, Dubey S, Flossmann O, Hall C, Hollywood J, Jayne D, Jones R, Lanyon P, Muir A, Scott D, Young L, Luqmani RA. Modification and validation of the Birmingham Vasculitis Activity Score (version 3). Ann Rheum Dis. 2009 Dec;68(12):1827-32. doi: 10.1136/ard.2008.101279. Epub 2008 Dec 3. PMID 19054820
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Rider LG, Koziol D, Giannini EH, Jain MS, Smith MR, Whitney-Mahoney K, Feldman BM, Wright SJ, Lindsley CB, Pachman LM, Villalba ML, Lovell DJ, Bowyer SL, Plotz PH, Miller FW, Hicks JE. Validation of manual muscle testing and a subset of eight muscles for adult and juvenile idiopathic inflammatory myopathies. Arthritis Care Res (Hoboken). 2010 Apr;62(4):465-72. doi: 10.1002/acr.20035. PMID 20391500
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Seror R, Ravaud P, Bowman SJ, Baron G, Tzioufas A, Theander E, Gottenberg JE, Bootsma H, Mariette X, Vitali C; EULAR Sjogren's Task Force. EULAR Sjogren's syndrome disease activity index: development of a consensus systemic disease activity index for primary Sjogren's syndrome. Ann Rheum Dis. 2010 Jun;69(6):1103-9. doi: 10.1136/ard.2009.110619. Epub 2009 Jun 28. PMID 19561361
- [Background] Stevens E, Weinblatt ME, Massarotti E, Griffin F, Emani S, Desai S. Safety of the Zoster Vaccine Recombinant Adjuvanted in Rheumatoid Arthritis and Other Systemic Rheumatic Disease Patients: A Single Center's Experience With 400 Patients. ACR Open Rheumatol. 2020 Jun;2(6):357-361. doi: 10.1002/acr2.11150. Epub 2020 May 15. PMID 32412669
- [Background] Tillett W, Costa L, Jadon D, Wallis D, Cavill C, McHugh J, Korendowych E, McHugh N. The ClASsification for Psoriatic ARthritis (CASPAR) criteria--a retrospective feasibility, sensitivity, and specificity study. J Rheumatol. 2012 Jan;39(1):154-6. doi: 10.3899/jrheum.110845. Epub 2011 Nov 15. PMID 22089469
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Background] Vink P, Delgado Mingorance I, Maximiano Alonso C, Rubio-Viqueira B, Jung KH, Rodriguez Moreno JF, Grande E, Marrupe Gonzalez D, Lowndes S, Puente J, Kristeleit H, Farrugia D, McNeil SA, Campora L, Di Paolo E, El Idrissi M, Godeaux O, Lopez-Fauqued M, Salaun B, Heineman TC, Oostvogels L; Zoster-028 Study Group. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine in patients with solid tumors, vaccinated before or during chemotherapy: A randomized trial. Cancer. 2019 Apr 15;125(8):1301-1312. doi: 10.1002/cncr.31909. Epub 2019 Feb 1. PMID 30707761
- [Background] Vink P, Ramon Torrell JM, Sanchez Fructuoso A, Kim SJ, Kim SI, Zaltzman J, Ortiz F, Campistol Plana JM, Fernandez Rodriguez AM, Rebollo Rodrigo H, Campins Marti M, Perez R, Gonzalez Roncero FM, Kumar D, Chiang YJ, Doucette K, Pipeleers L, Aguera Morales ML, Rodriguez-Ferrero ML, Secchi A, McNeil SA, Campora L, Di Paolo E, El Idrissi M, Lopez-Fauqued M, Salaun B, Heineman TC, Oostvogels L; Z-041 Study Group. Immunogenicity and Safety of the Adjuvanted Recombinant Zoster Vaccine in Chronically Immunosuppressed Adults Following Renal Transplant: A Phase 3, Randomized Clinical Trial. Clin Infect Dis. 2020 Jan 2;70(2):181-190. doi: 10.1093/cid/ciz177. PMID 30843046
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Wolfe F, Michaud K, Chakravarty EF. Rates and predictors of herpes zoster in patients with rheumatoid arthritis and non-inflammatory musculoskeletal disorders. Rheumatology (Oxford). 2006 Nov;45(11):1370-5. doi: 10.1093/rheumatology/kel328. Epub 2006 Sep 26. PMID 17003175
- [Background] Yun H, Yang S, Chen L, Xie F, Winthrop K, Baddley JW, Saag KG, Singh J, Curtis JR. Risk of Herpes Zoster in Autoimmune and Inflammatory Diseases: Implications for Vaccination. Arthritis Rheumatol. 2016 Sep;68(9):2328-37. doi: 10.1002/art.39670. PMID 26990731
- [Background] Criteria for diagnosis of Behcet's disease. International Study Group for Behcet's Disease. Lancet. 1990 May 5;335(8697):1078-80. PMID 1970380
- [Background] International Team for the Revision of the International Criteria for Behcet's Disease (ITR-ICBD). The International Criteria for Behcet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014 Mar;28(3):338-47. doi: 10.1111/jdv.12107. Epub 2013 Feb 26. PMID 23441863
- [Background] Petri M, Joyce D, Haag K, Fava A, Goldman DW, Zhong D, Xiao S, Milstone A, Magder LS. Effect of Systemic Lupus Erythematosus and Immunosuppressive Agents on COVID-19 Vaccination Antibody Response. Arthritis Care Res (Hoboken). 2023 Sep;75(9):1878-1885. doi: 10.1002/acr.25094. Epub 2023 Mar 1. PMID 36714913